CLINICAL TRIAL: NCT03239223
Title: A Randomised, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Evaluate Safety, Tolerability and Pharmacokinetics of Topical ABI-1968 in Subjects With Cervical High Grade Squamous Intreaepithelial Lesions (cHSIL)
Brief Title: Study of Topical ABI-1968 in Subjects With Precancerous Cervical Lesions From Human Papillomavirus (HPV) Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antiva Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ABI-1968-102
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: HSIL; HSIL of Cervix; High-Grade Squamous Intraepithelial Lesions; High-grade Cervical Intraepithelial Neoplasia; Human Papilloma Virus; Cervical Cancer; Cervical Intraepithelial Neoplasia; Cervical Neoplasm; Cervical Dysplasia; CIN
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: Up to two ascending dose cohorts (8 subjects per cohort) may receive multiple doses in 2 ascending dose strengths of ABI-1968 Topical Cream. After completing the multiple ascending dose portion a Cohort Expansion group of 32 to 40 subjects will be initiated.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose 1 - Multiple Ascending Dose (MAD) (Experimental): ABI-1968 or Placebo topical cream applied at Day 1, Day 8, Day 15 and Day 22
  Interventions: Drug: ABI-1968
- Dose 2 - Multiple Ascending Dose (MAD) (Experimental): ABI-1968 or Placebo topical cream applied at Day 1, Day 8, Day 15 and Day 22
  Interventions: Drug: ABI-1968

INTERVENTIONS:
Drug: ABI-1968 — Topical ABI-1968 Cream or Placebo with 4 doses administered up to 4 Cohorts

SUMMARY:
This study evaluates the use of topical ABI-1968 cream, in the treatment of cervical precancerous lesions in adult women.

ELIGIBILITY:
Inclusion Criteria:

* Women, 25 to 50 years old.
* Cervical HSIL diagnosis made within 2 months of enrollment and confirmed with biopsy with no evidence of invasive cancer in any specimen and must be p16+.
* Able and willing to abstain from sexual intercourse for 48 hours prior to first dose and 2 days after each dose.
* Generally experiencing regular menstrual cycles, unless using long-acting reversible contraception that induces amenorrhea (e.g., Mirena IUD, Norplant).

Exclusion Criteria:

* Women who are pregnant, plan to become pregnant in the next 4 months, or lactating females.
* History of cancer, except basal cell or squamous cell carcinoma of the skin.
* History of genital herpes with > 3 outbreaks per year, or active non-HPV vaginal infection.
* Plan to have excision or ablation of the lesion(s) within 3 months of enrollment.
* History of cervical cancer, colposcopy suspicious for cancer, any prior treatment of CIN, or hysterectomy.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of ABI-1968 for the treatment of cHSIL | 85 Days
  Number of participants with Adverse Events related to treatment to determine MTD

SECONDARY OUTCOMES:
Systemic exposure to Topical ABI-1968 Cream following topical application to the cervix. | 85 Days
  Plasma concentrations of ABI-1968 over time to determine systemic exposure
Histopathology of areas with biopsy-proven disease following multiple doses of Topical ABI-1968 Cream. | 85 Days
  Number of subjects with complete and or partial regression of cHSIL by Colposcopy and histopathology to determine change and impact over 4 weekly doses

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - Research Center, Los Angeles, California
  - Research Center, Lake Worth, Florida
  - Research Center, Idaho Falls, Idaho
  - Research Center, Chapel Hill, North Carolina
  - Research Center, Winston-Salem, North Carolina
  - Research Center, Norfolk, Virginia
- Australia (3):
  - Research Center, Camperdown, New South Wales
  - Research Center, Darlinghurst, New South Wales
  - Research Center, South Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No